CLINICAL TRIAL: NCT07343154
Title: A Prospective Study on the Effects of Percutaneous Patent Foramen Ovale Closure on Multimodal Brain Function, Cognition, and Emotion in Patients With Migraine and Patent Foramen Ovale
Brief Title: Multimodal Brain Function in Migraine Patients With Patent Foramen Ovale
Acronym: NEURO-PFO
Status: Not yet recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: LYEC2025-0277
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: PFO; Cognitive; Cognitive Functions; Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This investigator-initiated, single-center prospective study is designed to clarify how patent foramen ovale (PFO) relates to brain function abnormalities in patients with drug-refractory migraine with aura (MA), and whether percutaneous PFO closure is associated with measurable, longitudinal improvements in neurophysiological and neuroimaging markers as well as clinical symptoms.

The study addresses two core questions: (1) Do MA patients with clinically significant right-to-left shunt due to PFO demonstrate distinct resting-state brain function patterns-captured by high-density EEG (hdEEG), resting-state functional MRI (rs-fMRI), and standardized cognitive testing-compared with MA patients without PFO? (2) In MA patients with PFO who undergo clinically indicated percutaneous PFO closure, do these multimodal brain function measures change over time after closure (pre-procedure vs 1, 6, and 12 months), and are such changes accompanied by improvement in migraine burden, quality of life, and mood/anxiety symptoms? The protocol includes two phases. In Phase 1 (cross-sectional comparison), two groups are evaluated at baseline: MA with PFO (PFO+/MA+) and MA without PFO (PFO-/MA+). Participants complete hdEEG and rs-fMRI to characterize whole-brain power spectral density and connectivity, and undergo MATRICS Consensus Cognitive Battery (MCCB) testing and validated symptom/psychological assessments (e.g., MIDAS, MSQ v2.1, PHQ-9, GAD-7, RoPE). In Phase 2 (prospective self-controlled cohort), eligible PFO+/MA+ participants who proceed to percutaneous PFO closure as part of routine clinical care are followed longitudinally with repeated multimodal assessments at pre-closure baseline and post-closure 1, 6, and 12 months. This phase evaluates within-person trajectories of resting-state brain function (hdEEG, rs-fMRI) and cognition/emotion measures, together with migraine diary-based outcomes and patient-reported quality of life/disability and mood/anxiety scales. Key eligibility focuses on adults aged 18-65 years with ICHD-3-defined migraine with aura and a history of frequent migraine (≥4 migraine days/month during screening) despite prior preventive therapy trials; the PFO group requires echocardiographic confirmation of PFO with at least moderate right-to-left shunt (e.g., during Valsalva on contrast TEE), consistent with the study's focus on clinically meaningful shunt physiology.

The primary endpoints are multimodal brain function and cognition measures. In Phase 1, the main outcomes include between-group differences in MCCB composite score, rs-fMRI whole-brain functional connectivity strength, and hdEEG spectral power across frequency bands (delta/theta/alpha/beta/gamma) and theta-band connectivity quantified by whole-brain phase-lag index (PLI). In Phase 2, the primary outcome is the 12-month post-closure change in these multimodal resting-state brain function measures, reflecting dynamic neural recovery or reorganization after PFO closure.

Secondary outcomes include changes in migraine clinical metrics (monthly migraine days, attack frequency and duration, and complete remission rate), migraine-specific quality of life (MSQ v2.1), disability (MIDAS), and depression/anxiety symptom scores (PHQ-9 and GAD-7) over follow-up. Safety outcomes include adverse events potentially related to the closure procedure and routine post-procedural anti-thrombotic therapy, captured throughout follow-up.

DETAILED DESCRIPTION:
This is an investigator-initiated, single-center, prospective, longitudinal, self-controlled cohort study evaluating multimodal brain function changes in adults with migraine with aura and echocardiographically confirmed patent foramen ovale (PFO) who undergo clinically indicated percutaneous PFO closure as part of routine care. The study is designed to characterize within-person trajectories of resting-state neurophysiology, brain network organization, and neurocognitive performance from pre-closure baseline through post-closure follow-up, using standardized acquisition and analytic pipelines for high-density electroencephalography (hdEEG), resting-state functional MRI (rs-fMRI), and cognitive testing.

Overall design and clinical workflow integration

Participants are identified through routine clinical pathways (cardiology/structural heart disease and headache/neurology services). Study procedures are embedded within the standard pre-procedural assessment and post-procedural follow-up schedule whenever feasible to reduce participant burden and improve data completeness. The PFO closure procedure itself, device selection, peri-procedural management, and post-procedure antithrombotic therapy follow local clinical practice and are not assigned by the study.

Participants complete a pre-closure baseline assessment and then undergo repeated assessments during follow-up. Study visits are time-locked to clinically meaningful recovery phases after PFO closure and are intended to capture early neurophysiologic changes, intermediate adaptation, and longer-term stabilization of brain network measures.

Multimodal assessments and acquisition procedures Resting-state fMRI acquisition and quality control

Resting-state fMRI is acquired on a 3.0T clinical MRI system using standardized sequences suitable for network-level analyses. Participants are instructed to remain still, stay awake, and follow a uniform resting condition (e.g., eyes closed or eyes open with fixation) across all visits to maximize longitudinal comparability. Imaging quality control emphasizes minimization of head motion and physiological artifacts. Data are screened for completeness, scanner protocol deviations, and motion outliers; scans failing prespecified QC thresholds (e.g., excessive motion) are flagged for exclusion from network analyses, while retaining other usable outcomes when appropriate.

hdEEG acquisition and quality control

High-density EEG is recorded under standardized resting-state conditions. The acquisition protocol is harmonized across visits, including participant preparation, impedance checks, recording duration, and environment control (e.g., low-noise room, standardized instructions). Recording quality control includes monitoring for excessive muscle activity, eye movement contamination, channel artifacts, and drowsiness. Raw data are archived to enable reproducible preprocessing and re-analysis if needed.

Neurocognitive and symptom-related assessments

Neurocognitive performance is assessed using the MATRICS Consensus Cognitive Battery (MCCB) administered by trained staff following standardized procedures and scoring rules. Additional clinical assessments collected as part of the study support interpretation of multimodal brain measures over time (e.g., headache diary-derived metrics and validated patient-reported measures). These measures are collected with consistent timing relative to imaging/EEG when feasible to reduce measurement variability.

Neuroimaging and EEG preprocessing and network construction rs-fMRI preprocessing

Resting-state fMRI preprocessing follows established pipelines for connectome-based analyses, including: removal of initial volumes (if applicable), slice timing correction (if used), motion correction, coregistration to individual anatomical space (when available), normalization to standard space, nuisance regression (e.g., motion parameters; optionally physiological or WM/CSF signals depending on the finalized pipeline), temporal filtering, and spatial smoothing consistent with the selected atlas and connectivity approach. Motion is quantified using standard metrics (e.g., framewise displacement). Scrubbing/censoring strategies and sensitivity analyses (e.g., with/without global signal regression) may be applied to evaluate robustness.

hdEEG preprocessing

EEG preprocessing includes band-pass filtering, bad channel detection/interpolation, artifact attenuation (e.g., independent component analysis or equivalent methods to address ocular and muscle components), re-referencing strategy consistent with high-density recordings, and segmentation into resting epochs. Frequency-domain features (e.g., power spectral density in canonical bands) and connectivity measures are derived using standardized parameters across visits.

Parcellation (brain "atlas") and network generation

For rs-fMRI, the brain is parcellated into regions of interest (ROIs) using a predefined atlas (e.g., a functionally defined multi-network parcellation such as a Schaefer-based atlas, finalized prior to database lock). Regional time series are extracted per ROI and pairwise connectivity matrices are constructed using correlation-based metrics (with Fisher z-transformation where appropriate). For EEG, connectivity is computed using phase-based measures that reduce volume-conduction bias (e.g., phase-lag index-type metrics), with a focus on prespecified frequency bands relevant to resting-state network physiology. Network representations may include whole-brain connectivity matrices and derived within-network/between-network summaries aligned to canonical functional systems (e.g., default mode, salience, executive control networks), finalized a priori.

Statistical considerations and analysis approach (high level) Primary analytic framework

The primary analyses are within-person comparisons between pre-closure baseline and follow-up timepoints for multimodal brain function and cognition endpoints. Longitudinal modeling will be implemented using approaches appropriate for repeated measures, such as linear mixed-effects models with participant-specific random effects, allowing inclusion of all available timepoints and accommodating incomplete follow-up under a missing-at-random assumption. Time is modeled as categorical (visit-based) or continuous (time since closure) depending on the finalized specification.

Multiple primary endpoints and multiplicity control

Because the study includes two primary domains (neuroimaging/EEG-derived brain function and MCCB cognition), multiplicity control is applied to preserve the overall type I error rate. A Bonferroni-adjusted significance threshold is used for confirmatory testing across the two primary endpoints (i.e., α split across two primary tests). Secondary and exploratory analyses are interpreted with appropriate caution and are primarily hypothesis-generating.

Network-level inference and feature selection (exploratory components)

For connectome-wide rs-fMRI analyses, network-based inference methods (e.g., network-based statistics with permutation testing) may be used to identify subnetworks showing coherent changes across edges while controlling family-wise error at the component level. For EEG connectivity, analogous cluster-based or network-based permutation approaches may be used depending on the finalized feature set.

To relate multimodal network features to cognitive performance and clinical measures, multivariable modeling strategies may be applied. If the feature space is high-dimensional relative to sample size (e.g., edge-wise connectome features), regularization and feature-selection methods (e.g., LASSO or elastic net) can be used in an exploratory framework with cross-validation to reduce overfitting. Selected features can then be summarized (e.g., network strength indices) and examined for longitudinal association with MCCB change or symptom trajectories. These models are explicitly exploratory unless prespecified and adequately powered for prediction.

Covariates and confounding control

Models will consider key covariates that can influence brain network measures and cognition (e.g., age, sex, education, head motion metrics for fMRI, medication changes, and other clinically relevant factors). Sensitivity analyses may evaluate the impact of motion thresholds, preprocessing choices, and alternative atlas resolutions.

Missing data and data quality

Missingness may arise from loss to follow-up or unusable imaging/EEG data. The analysis plan prioritizes (1) preventing missing data through scheduling integration and QC feedback loops, and (2) transparent handling of missingness. Mixed-effects models enable inclusion of participants with partial follow-up, while imaging/EEG-specific QC exclusions are documented with reasons. Where applicable, sensitivity analyses will compare complete-case and all-available-data approaches.

Safety oversight and adverse event documentation

Although the study is non-interventional with respect to treatment assignment, it prospectively captures adverse events temporally associated with PFO closure and routine post-procedure management. Adverse events and serious adverse events are recorded throughout follow-up using standardized definitions, grading, attribution (e.g., procedure-related, device-related, medication-related, or unrelated), and reporting pathways consistent with institutional requirements. This safety documentation is observational and does not alter clinical management.

Data management, confidentiality, and reproducibility

Study data are recorded in a structured database with prespecified variable definitions and audit trails. Imaging and EEG data are stored in de-identified formats with controlled access. Data linkage between clinical records and research identifiers is maintained in a secured location accessible only to authorized personnel. Preprocessing pipelines, parameter settings, and analysis scripts are version-controlled to support reproducibility and transparent reporting.

Dissemination

Results will be disseminated through peer-reviewed publications and academic presentations. Reporting will follow relevant observational study guidelines and will distinguish prespecified confirmatory analyses from exploratory modeling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and <60 years at Screening/Baseline.
* Diagnosis of migraine with aura established by a neurologist according to the International Classification of Headache Disorders, 3rd edition (ICHD-3) criteria.
* Migraine history ≥1 year AND, during the 3-month screening/run-in period, an average of ≥4 migraine days per month; participant is willing and able to complete a headache diary, which will be reviewed by the investigator prior to enrollment.
* Patent foramen ovale (PFO) identified by transthoracic echocardiography (TTE) and confirmed by contrast transesophageal echocardiography (cTEE), with at least moderate atrial-level right-to-left shunt (RLS) during Valsalva maneuver.
* RLS grading by microbubbles in the left-sided cardiac chambers per frame on single-frame images:
* No RLS: 0 microbubbles
* Grade I (small): 1-10 microbubbles/frame
* Grade II (moderate): 11-30 microbubbles/frame
* Grade III (large): >30 microbubbles/frame or near-complete opacification of the left chambers ("hazy" appearance)
* Prior use of at least three different classes of migraine preventive therapies with either <50% improvement in migraine frequency during treatment OR intolerable adverse effects.
* At least two therapies must be from different categories among (a-f); the third may be one of (g-j):

  1. Beta-blockers
  2. Tricyclic antidepressants
  3. Verapamil or flunarizine
  4. Sodium valproate (or divalproex sodium)
  5. Topiramate
  6. Other anticonvulsants
  7. Any therapy supported as effective by at least one positive randomized controlled trial
  8. Nonsteroidal anti-inflammatory drugs (NSAIDs)
  9. Metabolic agents (e.g., vitamin B2 or coenzyme Q10)
  10. Traditional Chinese medicine
* Participant has been on a stable daily dose regimen of preventive headache medication for ≥3 consecutive months prior to enrollment (to be verified during screening).
* Written informed consent provided and willingness to comply with study procedures and follow-up schedule.

Exclusion Criteria:

* Expected life expectancy ≤1 year at Screening/Baseline.
* Secondary migraine attributable to other causes.
* History of transient ischemic attack (TIA), stroke, or intracranial hemorrhage.
* Investigator-determined anatomical findings on TEE that are unfavorable for successful PFO occluder deployment or any contraindication to device implantation, including (but not limited to):
* Inability to undergo/complete TEE
* Vascular access unable to accommodate the delivery system
* Requirement for transseptal puncture
* Requirement for implantation of more than one occluder
* Defect size estimated too large for successful closure
* Potential interference between the occluder and other intracardiac structures
* Anatomy preventing adequate apposition of the occluder discs to the atrial septum
* Allergy to any component/material of the AMPLATZER™ PFO Occluder (e.g., nickel allergy).
* Current or past diagnosis of severe psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depressive disorder), or unstable psychiatric illness defined as psychiatric hospitalization, medication dose adjustment, or marked symptom fluctuation within the past 6 months.
* Neurological and/or neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease, multiple sclerosis), uncontrolled epilepsy/seizures within the past 1 year, central nervous system tumor, or history of traumatic brain injury.
* History of myocardial infarction.
* History of pacemaker implantation, atrial septal defect (ASD) closure, or left atrial appendage (LAA) closure.
* Intracardiac right-to-left shunt due to causes other than PFO.
* Contraindications to aspirin and/or clopidogrel, including significant thrombocytopenia, major trauma, acute clinically significant bleeding, or allergy to study medications.
* Hepatic impairment defined as PT and/or APTT >2× the upper limit of normal (ULN) OR total bilirubin ≥3 mg/dL.
* Poorly controlled diabetes mellitus at Screening/Baseline (as judged by the investigator).
* Poorly controlled atrial fibrillation at Screening/Baseline (as judged by the investigator).
* Poorly controlled hypertension at Screening/Baseline, defined as blood pressure >160/90 mmHg despite appropriate pharmacologic treatment.
* Active autoimmune disease at Screening/Baseline (e.g., systemic lupus erythematosus, rheumatoid arthritis, polyarteritis nodosa, central nervous system granulomatous vasculitis).
* Active infection at Screening/Baseline that cannot be fully resolved prior to enrollment.
* Alcohol abuse or drug dependence at Screening/Baseline.
* Ongoing anticoagulation therapy that cannot be discontinued.
* Unable to accurately describe headache status and/or unable to complete/maintain a headache diary.
* Currently participating in another device or drug clinical trial in which the primary endpoint has not been reached, or that may clinically confound this study's endpoints, or that prohibits co-enrollment.
* Pregnant or planning pregnancy during the study period.
* Planned elective surgery during the study period.
* Any medical condition or circumstance that, in the investigator's opinion, poses a significant risk to participant safety, confounds study results, or interferes with study participation.
* Any other medical or non-medical reason that, in the investigator's opinion, makes the participant unsuitable (e.g., inability to comply with study procedures/visits, plans to relocate during the study period).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from the neurology headache clinic and structural heart/cardiology services at Xiangya 2nd hospital, a tertiary care teaching hospital in Changsha, China. Potential participants will be identified during routine clinical care among adults evaluated for migraine with aura and referred for echocardiographic assessment of suspected or known patent foramen ovale. Recruitment will occur in outpatient clinics and, when applicable, during inpatient admissions, with screening based on clinical diagnosis and standard-of-care imaging performed as part of usual practice.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in whole-brain network connectivity strength (FCN and MCN) from baseline to 12 months | from enrollment to the end of postoperative followup at 3 years
  Connectivity matrices will be constructed using a predefined brain parcellation; whole-brain connectivity strength will be summarized as a prespecified global network strength metric (and/or network-level strength within canonical systems).